CLINICAL TRIAL: NCT02393248
Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety and Tolerability Study of INCB054828 in Subjects With Advanced Malignancies (FIGHT-101)
Brief Title: Open-Label, Dose-Escalation Study of Pemigatinib in Subjects With Advanced Malignancies - (FIGHT-101)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-101
Expanded Access: NCT03906357 (No longer available)
Record Dates: First submitted 2015-01-30; First posted 2015-03-19 (Estimated); Results first posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Lung Cancer; Solid Tumor; Gastric Cancer; Urothelial Cancer; Endometrial Cancer; Multiple Myeloma; Myeloproliferative Neoplasms; Breast Cancer; Cholangiocarcinoma; UC; MPN
Keywords: alterations in FGF or FGFR; squamous non-small cell lung cancer; gastric cancer; urothelial cancer; endometrial cancer; multiple myeloma; MPN
MeSH Terms: conditions — Lung Neoplasms; Stomach Neoplasms; Endometrial Neoplasms; Multiple Myeloma; Myeloproliferative Disorders; Breast Neoplasms; Cholangiocarcinoma | interventions — pemigatinib; Gemcitabine; pembrolizumab; Docetaxel; Trastuzumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (25):
- Part 1: Intermittent pemigatinib 1/2/4 mg QD (Experimental): Participants self-administered oral pemigatinib 1/2/4 milligrams (mg) once daily (QD) on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
  Interventions: Drug: Pemigatinib
- Part 1: Intermittent pemigatinib 6 mg QD (Experimental): Participants self-administered oral pemigatinib 6 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
  Interventions: Drug: Pemigatinib
- Part 1: Intermittent pemigatinib 9 mg QD (Experimental): Participants self-administered oral pemigatinib 9 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
  Interventions: Drug: Pemigatinib
- Part 1: Intermittent pemigatinib 13.5 mg QD (Experimental): Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
  Interventions: Drug: Pemigatinib
- Part 1: Intermittent pemigatinib 20 mg QD (Experimental): Participants self-administered oral pemigatinib 20 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
  Interventions: Drug: Pemigatinib
- Part 1: Continuous pemigatinib 9 mg QD (Experimental): Participants self-administered oral pemigatinib 9 mg QD on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib
- Part 1: Continuous pemigatinib 13.5 mg QD (Experimental): Participants self-administered oral pemigatinib 13.5 mg QD on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib
- Part 1: Continuous pemigatinib 20 mg QD (Experimental): Participants self-administered oral pemigatinib 20 mg QD on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib
- Part 1: Continuous pemigatinib 7.5 mg BID (Experimental): Participants self-administered oral pemigatinib 7.5 mg twice daily (BID) on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib
- Part 1: Continuous pemigatinib 10 mg BID (Experimental): Participants self-administered oral pemigatinib 10 mg BID on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib
- Part 2: Intermittent pemigatinib 9 mg QD (Experimental): Participants self-administered oral pemigatinib 9 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
  Interventions: Drug: Pemigatinib
- Part 2: Intermittent pemigatinib 13.5 mg QD (Experimental): Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
  Interventions: Drug: Pemigatinib
- Part 2: Continuous pemigatinib 9 mg QD (Experimental): Participants self-administered oral pemigatinib 9 mg QD on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib
- Part 2: Continuous pemigatinib 13.5 mg QD (Experimental): Participants self-administered oral pemigatinib 13.5 mg QD on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib
- Part 2: Continuous pemigatinib 20 mg QD (Experimental): Participants self-administered oral pemigatinib 20 mg QD on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib
- Part 3: Gem/Cis/intermittent pemigatinib 9 mg (Experimental): Participants received gemcitabine (Gem) intravenously starting at 1000 mg/meters squared (m^2) (30 minutes) on Days 1 and 8 of each 21-day cycle. Cisplatin (Cis) was administered intravenously starting at 70 mg/m^2 (1-4 hours) once every 3 weeks on Day 1 of each 21-day cycle. Both gemcitabine and cisplatin doses could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued chemotherapy with medical monitor approval. Participants self-administered oral pemigatinib 9 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of gemcitabine/cisplatin.
  Interventions: Drug: Pemigatinib; Drug: Gemcitabine; Drug: Cisplatin
- Part 3: Gem/Cis/intermittent pemigatinib 13.5 mg (Experimental): Participants received gemcitabine intravenously starting at 1000 mg/m^2 (30 minutes) on Days 1 and 8 of each 21-day cycle. Cisplatin was administered intravenously starting at 70 mg/m^2 (1-4 hours) once every 3 weeks on Day 1 of each 21-day cycle. Both gemcitabine and cisplatin doses could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued chemotherapy with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of gemcitabine/cisplatin.
  Interventions: Drug: Pemigatinib; Drug: Gemcitabine; Drug: Cisplatin
- Part 3: Tras/intermittent pemigatinib 13.5 mg (Experimental): Trastuzumab (Tras) was administered as an open-label, commercial product at an initial dose of 8 mg/kilograms (kg) over a 90-minute intravenous infusion, followed by 6 mg/kg over a 30- to 90-minute intravenous infusion once every 3 weeks. The dose could have been adjusted for toxicity management, per commercial labeling. The investigator could have interrupted, modified, or discontinued trastuzumab with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of trastuzumab.
  Interventions: Drug: Pemigatinib; Drug: Trastuzumab
- Part 3: Doc/intermittent pemigatinib 13.5 mg (Experimental): Participants received docetaxel (Doc) intravenously starting at 75 mg/m^2 (1 hour) once every 3 weeks on Day 1 of each cycle. The dose could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued chemotherapy with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of docetaxel.
  Interventions: Drug: Pemigatinib; Drug: Docetaxel
- Part 3: Pem/intermittent pemigatinib 9 mg (Experimental): Participants received pembrolizumab (Pem) intravenously at 200 mg (30 minutes) once every 3 weeks on Day 1 of each cycle. The dose could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued pembrolizumab with medical monitor approval. Participants self-administered oral pemigatinib 9 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of pembrolizumab.
  Interventions: Drug: Pemigatinib; Drug: Pembrolizumab
- Part 3: Pem/intermittent pemigatinib 13.5 mg (Experimental): Participants received pembrolizumab intravenously at 200 mg (30 minutes) once every 3 weeks on Day 1 of each cycle. The dose could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued pembrolizumab with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of pembrolizumab.
  Interventions: Drug: Pemigatinib; Drug: Pembrolizumab
- Part 3: Pem/continuous pemigatinib 13.5 mg (Experimental): Participants received pembrolizumab intravenously at 200 mg (30 minutes) once every 3 weeks on Day 1 of each cycle. The dose could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued pembrolizumab with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on Days 1 through 21 of each 21-day cycle. It was permissible to continue pemigatinib administration during the toxicity break of pembrolizumab.
  Interventions: Drug: Pemigatinib; Drug: Pembrolizumab
- Part 3: Ref/continuous pemigatinib 9 mg (Experimental): Retifanlimab (Ref) was administered once every 4 weeks on a 28-day cycle as an open-label product, at an initial dose of 500 mg over a 60-minute intravenous infusion. Participants self-administered oral pemigatinib 9 mg QD on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib; Drug: Retifanlimab
- Part 3: Ref/continuous pemigatinib 13.5 mg (Experimental): Retifanlimab was administered once every 4 weeks on a 28-day cycle as an open-label product, at an initial dose of 500 mg over a 60-minute intravenous infusion. Participants self-administered oral pemigatinib 13.5 mg QD on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib; Drug: Retifanlimab
- Part 3: Ref/continuous pemigatinib 20 mg (Experimental): Retifanlimab was administered once every 4 weeks on a 28-day cycle as an open-label product, at an initial dose of 500 mg over a 60-minute intravenous infusion. Participants self-administered oral pemigatinib 20 mg QD on Days 1 through 21 of each 21-day cycle.
  Interventions: Drug: Pemigatinib; Drug: Retifanlimab

INTERVENTIONS:
Drug: Pemigatinib
  Other Names: INCB054828
Drug: Gemcitabine
  Arms: Part 3: Gem/Cis/intermittent pemigatinib 13.5 mg; Part 3: Gem/Cis/intermittent pemigatinib 9 mg
Drug: Pembrolizumab
  Arms: Part 3: Pem/continuous pemigatinib 13.5 mg; Part 3: Pem/intermittent pemigatinib 13.5 mg; Part 3: Pem/intermittent pemigatinib 9 mg
Drug: Docetaxel
  Arms: Part 3: Doc/intermittent pemigatinib 13.5 mg
Drug: Trastuzumab
  Arms: Part 3: Tras/intermittent pemigatinib 13.5 mg
Drug: Retifanlimab
  Other Names: INCMGA00012
  Arms: Part 3: Ref/continuous pemigatinib 13.5 mg; Part 3: Ref/continuous pemigatinib 20 mg; Part 3: Ref/continuous pemigatinib 9 mg
Drug: Cisplatin
  Arms: Part 3: Gem/Cis/intermittent pemigatinib 13.5 mg; Part 3: Gem/Cis/intermittent pemigatinib 9 mg

SUMMARY:
The purpose of this study will be to evaluate the safety, tolerability, and pharmacological activity of pemigatinib in subjects with advanced malignancies. This study will have three parts, dose escalation (Part 1), dose expansion (Part 2) and combination therapy (Part 3).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age 18 years or older on day of signing consent
2. Part 1: Any advanced solid tumor malignancy; Part 2: Subjects with squamous non-small cell lung cancer, cholangiocarcinoma/gastric cancer, urothelial cancer, breast/endometrial cancer, multiple myeloma, or MPNs that have a tumor or malignancy that has been evaluated and confirmed to harbor genetic alterations in FGF or FGFR genes. A subject's fibroblast growth factor (FGF) or fibroblast growth factor receptor (FGFR) alteration may be based on local or central laboratory results. Part 3: Dose finding: subjects with solid tumor malignancies who qualify for combo therapy; dose-expansion: FGF/FGFR+ subjects qualified to receive combo therapy
3. Has progressed after prior therapy and there is no further effective standard anticancer therapy available (including subject refuses or is intolerant)
4. Life expectancy > 12 weeks
5. Eastern Cooperative Oncology Group (ECOG) performance status:

   * Part 1: 0 or 1
   * Part 2 and 3: 0, 1, or 2

Exclusion Criteria:

1. Treatment with other investigational study drug for any indication for any reason, or receipt of anticancer medications within 21 days or 5 half-lives before first dose of study drug
2. Prior receipt of a selective FGFR inhibitor
3. History of a calcium/phosphate homeostasis disorder
4. History and/or current evidence of ectopic mineralization/calcification
5. Current evidence of corneal disorder/keratopathy
6. Has a history or presence of inadequate liver, renal, hematopoietic and/or cardiac function parameters outside protocol-defined range
7. Prior radiotherapy within 2 weeks of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Féliz, MD, Study Director — Incyte Corporation
Locations (20):
- United States (19):
  - University of Alabama At Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Cedars-Sinai Medical Center, West Hollywood, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Hematology Oncology Associates of the Tr, Port Saint Lucie, Florida
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Northwell Health - Monter Cancer Center, New Hyde Park, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University - Wexner Medical Center, Columbus, Ohio
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - Mary Crowley Cancer Research Ctr, Dallas, Texas
  - Md Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Baylor Scott & White Health, Temple, Texas
- The Finsen Centre National Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Subbiah V, Iannotti NO, Gutierrez M, Smith DC, Feliz L, Lihou CF, Tian C, Silverman IM, Ji T, Saleh M. FIGHT-101, a first-in-human study of potent and selective FGFR 1-3 inhibitor pemigatinib in pan-cancer patients with FGF/FGFR alterations and advanced malignancies. Ann Oncol. 2022 May;33(5):522-533. doi: 10.1016/j.annonc.2022.02.001. Epub 2022 Feb 14. PMID 35176457
- [Derived] Gong X, Ji T, Liu X, Chen X, Yeleswaram S. Evaluation of the clinical cardiac safety of pemigatinib, a fibroblast growth factor receptor inhibitor, in participants with advanced malignancies. Pharmacol Res Perspect. 2022 Feb;10(1):e00906. doi: 10.1002/prp2.906. PMID 34951522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 15 study sites: 14 sites in the United States and 1 site in Denmark. The study was conducted in 3 parts. Participants self-administered once daily doses of pemigatinib on a 2-weeks-on/1-week-off therapy (intermittent) or continuous schedule in 21-day cycles. Participants also self-administered twice daily doses of pemigatinib on a continuous schedule.
Groups:
- Part 3: Gem/Cis/Intermittent Pemigatinib 9 mg: Participants received gemcitabine (Gem) intravenously starting at 1000 mg/meters squared (m^2) on Days 1 and 8 of each 21-day cycle. Cisplatin (Cis) was administered intravenously starting at 70 mg/m^2 once every 3 weeks on Day 1 of each 21-day cycle. Both gemcitabine and cisplatin doses could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued chemotherapy with medical monitor approval. Participants self-administered oral pemigatinib 9 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of gemcitabine/cisplatin.
- Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg: Participants received gemcitabine intravenously starting at 1000 mg/m^2 on Days 1 and 8 of each 21-day cycle. Cisplatin was administered intravenously starting at 70 mg/m^2 once every 3 weeks on Day 1 of each 21-day cycle. Both gemcitabine and cisplatin doses could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued chemotherapy with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of gemcitabine/cisplatin.
- Part 3: Tras/Intermittent Pemigatinib 13.5 mg: Trastuzumab (Tras) was administered as an open-label, commercial product at an initial intravenous dose of 8 mg/kilograms (kg), followed by 6 mg/kg intravenously once every 3 weeks. The dose could have been adjusted for toxicity management, per commercial labeling. The investigator could have interrupted, modified, or discontinued trastuzumab with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of trastuzumab.
- Part 3: Doc/Intermittent Pemigatinib 13.5 mg: Participants received docetaxel (Doc) intravenously starting at 75 mg/m^2 once every 3 weeks on Day 1 of each cycle. The dose could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued chemotherapy with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of docetaxel.
- Part 3: Pem/Intermittent Pemigatinib 9 mg: Participants received pembrolizumab (Pem) intravenously at 200 mg once every 3 weeks on Day 1 of each cycle. The dose could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued pembrolizumab with medical monitor approval. Participants self-administered oral pemigatinib 9 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of pembrolizumab.
- Part 3: Pem/Intermittent Pemigatinib 13.5 mg: Participants received pembrolizumab intravenously at 200 mg once every 3 weeks on Day 1 of each cycle. The dose could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued pembrolizumab with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. It was permissible to continue pemigatinib administration during the toxicity break of pembrolizumab.
- Part 3: Pem/Continuous Pemigatinib 13.5 mg: Participants received pembrolizumab intravenously at 200 mg once every 3 weeks on Day 1 of each cycle. The dose could have been adjusted for toxicity management per commercial labeling. The investigator could have interrupted, modified, or discontinued pembrolizumab with medical monitor approval. Participants self-administered oral pemigatinib 13.5 mg QD on Days 1 through 21 of each 21-day cycle. It was permissible to continue pemigatinib administration during the toxicity break of pembrolizumab.
- Part 3: Ref/Continuous Pemigatinib 9 mg: Retifanlimab (Ref) was administered once every 4 weeks on a 28-day cycle as an open-label product, at an initial intravenous dose of 500 mg. Participants self-administered oral pemigatinib 9 mg QD on Days 1 through 21 of each 21-day cycle.
- Part 3: Ref/Continuous Pemigatinib 13.5 mg: Retifanlimab was administered once every 4 weeks on a 28-day cycle as an open-label product, at an initial intravenous dose of 500 mg. Participants self-administered oral pemigatinib 13.5 mg QD on Days 1 through 21 of each 21-day cycle.
- Part 3: Ref/Continuous Pemigatinib 20 mg: Retifanlimab was administered once every 4 weeks on a 28-day cycle as an open-label product, at an initial intravenous dose of 500 mg. Participants self-administered oral pemigatinib 20 mg QD on Days 1 through 21 of each 21-day cycle.
Period: Part 1: Monotherapy Dose Escalation
Arm/Group | Part 1: Intermittent Pemigatinib 1/2/4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Part 1: Intermittent Pemigatinib 9 mg QD | Part 1: Intermittent Pemigatinib 13.5 mg QD | Part 1: Intermittent Pemigatinib 20 mg QD | Part 1: Continuous Pemigatinib 9 mg QD | Part 1: Continuous Pemigatinib 13.5 mg QD | Part 1: Continuous Pemigatinib 20 mg QD | Part 1: Continuous Pemigatinib 7.5 mg BID | Part 1: Continuous Pemigatinib 10 mg BID | Part 2: Intermittent Pemigatinib 9 mg QD | Part 2: Intermittent Pemigatinib 13.5 mg QD | Part 2: Continuous Pemigatinib 9 mg QD | Part 2: Continuous Pemigatinib 13.5 mg QD | Part 2: Continuous Pemigatinib 20 mg QD | Part 3: Gem/Cis/Intermittent Pemigatinib 9 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 9 mg | Part 3: Ref/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 20 mg
Started | 3 | 4 | 3 | 6 | 6 | 9 | 10 | 9 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 3 | 6 | 6 | 9 | 9 | 8 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 3 | 6 | 6 | 6 | 5 | 8 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Decline; Withdrew by Physician | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Monotherapy Dose Expansion
Arm/Group | Part 1: Intermittent Pemigatinib 1/2/4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Part 1: Intermittent Pemigatinib 9 mg QD | Part 1: Intermittent Pemigatinib 13.5 mg QD | Part 1: Intermittent Pemigatinib 20 mg QD | Part 1: Continuous Pemigatinib 9 mg QD | Part 1: Continuous Pemigatinib 13.5 mg QD | Part 1: Continuous Pemigatinib 20 mg QD | Part 1: Continuous Pemigatinib 7.5 mg BID | Part 1: Continuous Pemigatinib 10 mg BID | Part 2: Intermittent Pemigatinib 9 mg QD | Part 2: Intermittent Pemigatinib 13.5 mg QD | Part 2: Continuous Pemigatinib 9 mg QD | Part 2: Continuous Pemigatinib 13.5 mg QD | Part 2: Continuous Pemigatinib 20 mg QD | Part 3: Gem/Cis/Intermittent Pemigatinib 9 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 9 mg | Part 3: Ref/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 20 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 44 | 5 | 20 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 44 | 5 | 20 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 29 | 4 | 15 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3: Combination Therapy
Arm/Group | Part 1: Intermittent Pemigatinib 1/2/4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Part 1: Intermittent Pemigatinib 9 mg QD | Part 1: Intermittent Pemigatinib 13.5 mg QD | Part 1: Intermittent Pemigatinib 20 mg QD | Part 1: Continuous Pemigatinib 9 mg QD | Part 1: Continuous Pemigatinib 13.5 mg QD | Part 1: Continuous Pemigatinib 20 mg QD | Part 1: Continuous Pemigatinib 7.5 mg BID | Part 1: Continuous Pemigatinib 10 mg BID | Part 2: Intermittent Pemigatinib 9 mg QD | Part 2: Intermittent Pemigatinib 13.5 mg QD | Part 2: Continuous Pemigatinib 9 mg QD | Part 2: Continuous Pemigatinib 13.5 mg QD | Part 2: Continuous Pemigatinib 20 mg QD | Part 3: Gem/Cis/Intermittent Pemigatinib 9 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 9 mg | Part 3: Ref/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 20 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 6 | 7 | 3 | 14 | 9 | 7 | 9 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 6 | 7 | 3 | 14 | 9 | 7 | 8 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 5 | 5 | 3 | 7 | 5 | 6 | 3 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 1
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Rolled Over to Another Protocol after Receiving Same Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Placed on Hospice; Declined Further Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Intermittent Pemigatinib 1/2/4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Part 1: Intermittent Pemigatinib 9 mg QD | Part 1: Intermittent Pemigatinib 13.5 mg QD | Part 1: Intermittent Pemigatinib 20 mg QD | Part 1: Continuous Pemigatinib 9 mg QD | Part 1: Continuous Pemigatinib 13.5 mg QD | Part 1: Continuous Pemigatinib 20 mg QD | Part 1: Continuous Pemigatinib 7.5 mg BID | Part 1: Continuous Pemigatinib 10 mg BID | Part 2: Intermittent Pemigatinib 9 mg QD | Part 2: Intermittent Pemigatinib 13.5 mg QD | Part 2: Continuous Pemigatinib 9 mg QD | Part 2: Continuous Pemigatinib 13.5 mg QD | Part 2: Continuous Pemigatinib 20 mg QD | Part 3: Gem/Cis/Intermittent Pemigatinib 9 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 9 mg | Part 3: Ref/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 20 mg | Total
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 6 | 9 | 10 | 9 | 4 | 3 | 4 | 44 | 5 | 20 | 6 | 1 | 7 | 6 | 7 | 3 | 14 | 9 | 7 | 9 | 2 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (11.24) | 45.5 (17.31) | 56.3 (4.93) | 59.0 (14.79) | 56.2 (11.89) | 57.9 (15.70) | 61.2 (16.88) | 56.3 (15.19) | 66.8 (4.57) | 68.7 (15.89) | 50.3 (12.39) | 57.7 (11.81) | 63.8 (10.69) | 57.4 (13.78) | 58.3 (8.80) | 61.0 (NA) — The standard deviation was not calculated for a single participant. | 54.1 (10.43) | 47.8 (14.44) | 62.4 (9.16) | 55.0 (15.72) | 64.7 (10.50) | 61.8 (10.89) | 63.4 (11.43) | 66.9 (8.80) | 68.0 (7.07) | 59.0 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 3 | 3 | 6 | 5 | 6 | 0 | 2 | 3 | 27 | 5 | 10 | 5 | 0 | 3 | 4 | 3 | 1 | 5 | 3 | 7 | 5 | 1 | 113
  Male | 1 | 2 | 1 | 3 | 3 | 3 | 5 | 3 | 4 | 1 | 1 | 17 | 0 | 10 | 1 | 1 | 4 | 2 | 4 | 2 | 9 | 6 | 0 | 4 | 1 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 15
  Not Hispanic or Latino | 2 | 3 | 3 | 6 | 4 | 8 | 9 | 9 | 4 | 3 | 3 | 39 | 5 | 16 | 6 | 1 | 7 | 6 | 7 | 3 | 13 | 8 | 7 | 9 | 1 | 182
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 3 | 4 | 2 | 6 | 5 | 8 | 10 | 8 | 4 | 3 | 3 | 37 | 5 | 18 | 6 | 1 | 5 | 6 | 6 | 2 | 10 | 9 | 7 | 9 | 1 | 178
  Black/African-American | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 15
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  American-Indian/Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Captured as Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Parts 1 and 2 Combined: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: Adverse events were defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occurred after a participant provided informed consent. Abnormal laboratory values or test results that occurred after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). TEAEs were defined as adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug and within 30 days of the last dose of study drug.
Time Frame: up to 763 days
Population: Safety Population: all enrolled participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Intermittent Pemigatinib 1/2/4 mg QD: Participants self-administered oral pemigatinib 1/2/4 milligrams (mg) once daily (QD) on a 2-weeks-on therapy and 1-week-off therapy schedule in Part 1. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
- Part 1: Intermittent Pemigatinib 6 mg QD: Participants self-administered oral pemigatinib 6 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule in Part 1. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
- Parts 1 and 2: Intermittent Pemigatinib 9 mg QD: Participants self-administered oral pemigatinib 9 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule in either Part 1 or Part 2. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
- Parts 1 and 2: Intermittent Pemigatinib 13.5 mg QD: Participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule in either Part 1 or Part 2. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
- Part 1: Intermittent Pemigatinib 20 mg QD: Participants self-administered oral pemigatinib 20 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule in Part 1. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
- Parts 1 and 2: Continuous Pemigatinib 9 mg QD: Participants self-administered oral pemigatinib 9 mg QD on Days 1 through 21 of each 21-day cycle in either Part 1 or Part 2.
- Parts 1 and 2: Continuous Pemigatinib 13.5 mg QD: Participants self-administered oral pemigatinib 13.5 mg QD on Days 1 through 21 of each 21-day cycle in either Part 1 or Part 2.
- Parts 1 and 2: Continuous Pemigatinib 20 mg QD: Participants self-administered oral pemigatinib 20 mg QD on Days 1 through 21 of each 21-day cycle in either Part 1 or Part 2.
Arm/Group | Part 1: Intermittent Pemigatinib 1/2/4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent Pemigatinib 13.5 mg QD | Part 1: Intermittent Pemigatinib 20 mg QD | Parts 1 and 2: Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Continuous Pemigatinib 20 mg QD | Part 1: Continuous Pemigatinib 7.5 mg BID | Part 1: Continuous Pemigatinib 10 mg BID
Number analyzed (Participants) | 3 | 4 | 7 | 50 | 6 | 14 | 30 | 15 | 4 | 3
Participants | 3 | 3 | 7 | 50 | 6 | 14 | 30 | 15 | 4 | 3

2. Primary Outcome: Part 3: Number of Participants With Any TEAE
Description: as for outcome 1
Time Frame: up to 869 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: Gem/Cis/Intermittent Pemigatinib 9 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 9 mg | Part 3: Ref/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 20 mg
Number analyzed (Participants) | 1 | 7 | 6 | 7 | 3 | 14 | 9 | 7 | 9 | 2
Participants | 1 | 7 | 6 | 7 | 3 | 14 | 9 | 7 | 9 | 2

3. Primary Outcome: E0 Following Once Daily Dosing of Pemigatinib as Monotherapy in Parts 1 and 2
Description: E0 was defined as the Baseline serum concentration of phosphate.
Time Frame: predose on Days 1 and 14 of Cycle 1; anytime during visit on Day 1 of Cycle 2 and all subsequent cycles
Population: Pharmacokinetic/Pharmacodynamic (PK/PD) Population: all enrolled participants who had PK/PD data. The average serum concentration of phosphate on Cycle 1 Days 8 and 15 was chosen as a dependent variable for E-R analysis, which was independent of the intermittent dosing and continuous dosing regimens. Therefore, the intermittent dosing and continuous dosing groups from Parts 1 and 2 were combined into a single analysis group for E-R analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per deciliter (mg/dL)
Groups:
- Parts 1 and 2: Intermittent or Continuous Pemigatinib: Participant self-administered intermittent pemigatinib once daily (QD) or continuous pemigatinib QD or twice daily (BID). Intermittent dosing: participants self-administered oral pemigatinib 1/2/4 milligrams (mg), 6 mg, 9 mg, 13.5 mg, or 20 mg once daily (QD) on a 2-weeks-on therapy and 1-week-off therapy schedule in Part 1 or Part 2. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. Continuous dosing: participants self-administered oral pemigatinib 9 mg, 13.5 mg, or 20 mg QD on Days 1 through 21 of each 21-day cycle in Part 1 or Part 2. Participants self-administered oral pemigatinib 7.5 mg or 10 mg BID on Days 1 through 21 of each 21-day cycle in Part 1.
Arm/Group | Parts 1 and 2: Intermittent or Continuous Pemigatinib
Number analyzed (Participants) | 93
milligrams per deciliter (mg/dL) | 3.66 (1.91)

4. Primary Outcome: EC50 Following Once Daily Dosing of Pemigatinib as Monotherapy in Parts 1 and 2
Description: EC50 was defined as the pemigatinib steady-state area under the plasma or serum concentration-time curve that increases 50% of serum phosphate.
Time Frame: predose on Days 1 and 14 of Cycle 1; anytime during visit on Day 1 of Cycle 2 and all subsequent cycles
Population: PK/PD Population. The average serum concentration of phosphate on Cycle 1 Days 8 and 15 was chosen as a dependent variable for E-R analysis, which was independent of the intermittent dosing and continuous dosing regimens. Therefore, the intermittent dosing and continuous dosing groups from Parts 1 and 2 were combined into a single analysis group for E-R analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomoles
Arm/Group | Parts 1 and 2: Intermittent or Continuous Pemigatinib
Number analyzed (Participants) | 93
hours*nanomoles | 1573 (21.6)

5. Primary Outcome: Emax Following Once Daily Dosing of Pemigatinib as Monotherapy in Parts 1 and 2
Description: Emax was defined as the maximum degree of increasing of serum phosphate by pemigatinib.
Time Frame: predose on Days 1 and 14 of Cycle 1; anytime during visit on Day 1 of Cycle 2 and all subsequent cycles
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | Parts 1 and 2: Intermittent or Continuous Pemigatinib
Number analyzed (Participants) | 93
mg/dL | 5.76 (7.76)

6. Primary Outcome: Highest Serum Phosphate Concentration Following Pemigatinib as Monotherapy in Parts 1 and 2
Description: Serum phosphate concentration was assessed throughout Parts 1 and 2.
Time Frame: predose on Days 1 and 14 of Cycle 1; anytime during visit on Day 1 of Cycle 2 and all subsequent cycles
Population: as for outcome 4
Measure: Number; unit: mg/dL
Arm/Group | Parts 1 and 2: Intermittent or Continuous Pemigatinib
Number analyzed (Participants) | 93
mg/dL
  Minimum value in range of highest values for all participants | 3.5
  Maximum value in range of highest values for all participants | 11.2

7. Secondary Outcome: Part 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, as determined by the investigator. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 126 days
Population: Efficacy Evaluable Population: all enrolled participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Intermittent Pemigatinib 9 mg QD | Part 2: Intermittent Pemigatinib 13.5 mg QD | Part 2: Continuous Pemigatinib 9 mg QD | Part 2: Continuous Pemigatinib 13.5 mg QD | Part 2: Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 4 | 44 | 5 | 20 | 6
percentage of participants | 25.0 [0.6 to 80.6] | 4.5 [0.6 to 15.5] | 0.0 [0.0 to 52.2] | 30.0 [11.9 to 54.3] | 0.0 [0.0 to 45.9]

8. Secondary Outcome: Part 3: ORR
Description: ORR was defined as the percentage of participants with a best overall response of CR or PR, per RECIST version 1.1, as determined by the investigator. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 203 days
Population: Efficacy Evaluable Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3: Gem/Cis/Intermittent Pemigatinib 9 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 9 mg | Part 3: Ref/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 20 mg
Number analyzed (Participants) | 1 | 7 | 6 | 7 | 3 | 14 | 9 | 7 | 9 | 2
percentage of participants | 0.0 [0.0 to 97.5] | 42.9 [9.9 to 81.6] | 0.0 [0.0 to 45.9] | 14.3 [0.4 to 57.9] | 0.0 [0.0 to 70.8] | 28.6 [8.4 to 58.1] | 33.3 [7.5 to 70.1] | 0.0 [0.0 to 41.0] | 22.2 [2.8 to 60.0] | 0.0 [0.0 to 84.2]

9. Secondary Outcome: Parts 1 and 2: Cmax After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Day 1
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: Part 1: predose; 0.5, 1, 2, 4, 6, and 8 hours post-dose post-dose on Cycle 1 Day 1. Part 2: predose on Cycle 1 Day 1
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part 1: Intermittent Pemigatinib 1 mg QD: Participants self-administered oral pemigatinib 1 milligram (mg) once daily (QD) on a 2-weeks-on therapy and 1-week-off therapy schedule in Part 1. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
- Part 1: Intermittent Pemigatinib 2 mg QD: Participants self-administered oral pemigatinib 2 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule in Part 1. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
- Part 1: Intermittent Pemigatinib 4 mg QD: Participants self-administered oral pemigatinib 4 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule in Part 1. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break.
- Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD: Participants self-administered intermittent or continuous oral pemigatinib 9 mg QD in either Part 1 or Part 2. Intermittent dosing: participants self-administered oral pemigatinib 9 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule in either Part 1 or Part 2. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. Continuous dosing: participants self-administered oral pemigatinib 9 mg QD on Days 1 through 21 of each 21-day cycle in either Part 1 or Part 2.
- Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD: Participants self-administered intermittent or continuous oral pemigatinib 13.5 mg QD in either Part 1 or Part 2. Intermittent dosing: participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule in either Part 1 or Part 2. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. Continuous dosing: participants self-administered oral pemigatinib 13.5 mg QD on Days 1 through 21 of each 21-day cycle in either Part 1 or Part 2.
- Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD: Participants self-administered intermittent or continuous oral pemigatinib 20 mg QD in either Part 1 or Part 2. Intermittent dosing: participants self-administered oral pemigatinib 20 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule in Part 1. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. Continuous dosing: participants self-administered oral pemigatinib 20 mg QD on Days 1 through 21 of each 21-day cycle in either Part 1 or Part 2.
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 21 | 69 | 69
nanograms per milliliter (ng/mL) | 25.3 (NA) — A standard deviation was not calculated for a single participant. | 13.6 (NA) — A standard deviation was not calculated for a single participant. | 109 (NA) — A standard deviation was not calculated for a single participant. | 64.6 (9.16) | 139 (79.8) | 196 (121) | 300 (135)

10. Secondary Outcome: Parts 1 and 2: Tmax After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Day 1
Description: tmax was defined as the time to the maximum observed plasma concentration.
Time Frame: Part 1: predose; 0.5, 1, 2, 4, 6, and 8 hours post-dose post-dose on Cycle 1 Day 1. Part 2: predose on Cycle 1 Day 1
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 21 | 69 | 69
hours (hr) | 1 [NA to NA] — A range was not available for a single participant. | 5.92 [NA to NA] — A range was not available for a single participant. | 2.02 [NA to NA] — A range was not available for a single participant. | 1.14 [1.00 to 2.08] | 1.17 [0.500 to 2.13] | 1.20 [0.400 to 26.1] | 1.98 [0.500 to 22.9]

11. Secondary Outcome: Parts 1 and 2: AUClast After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Day 1
Description: AUClast was defined as the area under the plasma or serum concentration-time curve from the time of dosing to the last measurable concentration.
Time Frame: Part 1: predose; 0.5, 1, 2, 4, 6, and 8 hours post-dose post-dose on Cycle 1 Day 1. Part 2: predose on Cycle 1 Day 1
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 21 | 69 | 69
hr*ng/mL | 190 (NA) — A standard deviation was not calculated for a single participant. | 68.8 (NA) — A standard deviation was not calculated for a single participant. | 1010 (NA) — A standard deviation was not calculated for a single participant. | 641 (116) | 1140 (498) | 1820 (1210) | 2510 (935)

12. Secondary Outcome: Parts 1 and 2: AUC0-24 After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Day 1
Description: AUC0-24 was defined as the area under the plasma or serum concentration-time curve from time 0 to 24 hours post-dose.
Time Frame: Part 1: predose; 0.5, 1, 2, 4, 6, and 8 hours post-dose post-dose on Cycle 1 Day 1. Part 2: predose on Cycle 1 Day 1
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 21 | 69 | 69
hr*ng/mL | 191 (NA) — A standard deviation was not calculated for a single participant. | NA (NA) — A standard deviation was not calculated for a single participant. | 1010 (NA) — A standard deviation was not calculated for a single participant. | 644 (115) | 1150 (497) | 1840 (1080) | 2850 (1050)

13. Secondary Outcome: Parts 1 and 2: Cmax After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Days 8 and 14 (Steady State)
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: Part 1: predose on Cycle 1 Days 8 and 14; 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 14. Part 2: predose on Cycle 1 Days 8 and 14; 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 14
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 18 | 57 | 13
ng/mL | 26.2 (NA) — A standard deviation was not calculated for a single participant. | 22.9 (NA) — A standard deviation was not calculated for a single participant. | 103 (NA) — A standard deviation was not calculated for a single participant. | 86.1 (38.0) | 196 (123) | 271 (151) | 449 (172)
Statistical Analysis 1: Comparison: Part 1: Intermittent Pemigatinib 6 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD; Test type: Superiority; p = 0.2841, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 2: Comparison: Part 1: Intermittent Pemigatinib 6 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD; Test type: Superiority; p = 0.3042, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 3: Comparison: Part 1: Intermittent Pemigatinib 6 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD; Test type: Superiority; p = 0.1259, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 4: Comparison: Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD; Test type: Superiority; p = 0.8214, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 5: Comparison: Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD; Test type: Superiority; p = 0.4315, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 6: Comparison: Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD; Test type: Superiority; p = 0.2595, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)

14. Secondary Outcome: Parts 1 and 2: Tmax After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Days 8 and 14 (Steady State)
Description: tmax was defined as the time to the maximum observed plasma concentration.
Time Frame: as for outcome 13
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: hr
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 18 | 57 | 13
hr | 1.07 [NA to NA] — A range was not available for a single participant. | 3.98 [NA to NA] — A range was not available for a single participant. | 2.02 [NA to NA] — A range was not available for a single participant. | 1.58 [0.983 to 23.7] | 1.00 [0.500 to 6.10] | 1.13 [0.500 to 6.00] | 1.12 [0.517 to 5.90]

15. Secondary Outcome: Parts 1 and 2: t1/2 After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Days 8 and 14 (Steady State)
Description: t1/2 was defined as the apparent plasma terminal phase disposition half-life.
Time Frame: as for outcome 13
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 18 | 57 | 13
hr | 10.9 (NA) — A standard deviation was not calculated for a single participant. | 18.1 (NA) — A standard deviation was not calculated for a single participant. | 30.4 (NA) — A standard deviation was not calculated for a single participant. | 21.0 (22.8) | 17.2 (9.70) | 17.4 (9.64) | 13.1 (6.01)

16. Secondary Outcome: Parts 1 and 2: Cmin After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Days 8 and 14 (Steady State)
Description: Cmin was defined as the minimum observed plasma concentration over the dose interval.
Time Frame: as for outcome 13
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 18 | 57 | 13
ng/mL | 3.24 (NA) — A standard deviation was not calculated for a single participant. | 7.87 (NA) — A standard deviation was not calculated for a single participant. | 23.9 (NA) — A standard deviation was not calculated for a single participant. | 30.0 (15.1) | 49.9 (49.6) | 71.7 (56.7) | 104 (93.3)

17. Secondary Outcome: Parts 1 and 2: AUC0-24 After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Days 8 and 14 (Steady State)
Description: AUC0-24 was defined as the area under the plasma or serum concentration-time curve from time 0 to 24 hours post-dose.
Time Frame: as for outcome 13
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 18 | 57 | 13
hr*ng/mL | 208 (NA) — A standard deviation was not calculated for a single participant. | 322 (NA) — A standard deviation was not calculated for a single participant. | 1380 (NA) — A standard deviation was not calculated for a single participant. | 1080 (301) | 2180 (1630) | 3010 (1890) | 4350 (1480)
Statistical Analysis 1: Comparison: Part 1: Intermittent Pemigatinib 6 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD; Test type: Superiority; p = 0.8577, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 2: Comparison: Part 1: Intermittent Pemigatinib 6 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD; Test type: Superiority; p = 0.7238, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 3: Comparison: Part 1: Intermittent Pemigatinib 6 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD; Test type: Superiority; p = 0.5923, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 4: Comparison: Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD; Test type: Superiority; p = 0.7634, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 5: Comparison: Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD; Test type: Superiority; p = 0.5749, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)
Statistical Analysis 6: Comparison: Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD vs Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD; Test type: Superiority; p = 0.6877, ANOVA; 1-factor ANOVA of log-transformed, dose-normalized data (factor = dose)

18. Secondary Outcome: Parts 1 and 2: CL/F After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Days 8 and 14 (Steady State)
Description: CL/F was defined as the apparent oral dose clearance.
Time Frame: as for outcome 13
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Liters per hr (L/hr)
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 18 | 57 | 13
Liters per hr (L/hr) | 9.86 (NA) — A standard deviation was not calculated for a single participant. | 12.8 (NA) — A standard deviation was not calculated for a single participant. | 5.93 (NA) — A standard deviation was not calculated for a single participant. | 12.0 (3.14) | 15.7 (17.7) | 11.9 (5.72) | 10.3 (3.01)

19. Secondary Outcome: Parts 1 and 2: Vz/F After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Days 8 and 14 (Steady State)
Description: Vz/F was defined as the apparent volume of distribution.
Time Frame: as for outcome 13
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 18 | 57 | 13
Liters | 156 (NA) — A standard deviation was not calculated for a single participant. | 334 (NA) — A standard deviation was not calculated for a single participant. | 260 (NA) — A standard deviation was not calculated for a single participant. | 301 (241) | 246 (76.1) | 274 (165) | 180 (49.1)

20. Secondary Outcome: Parts 1 and 2: Accumulation Ratio After Once Daily Dosing of Pemigatinib as Monotherapy on Cycle 1 Days 8 and 14 (Steady State)
Description: The accumulation ratio was defined as the ratio of the accumulation of a drug under steady-state conditions as compared to a single dose.
Time Frame: as for outcome 13
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1: Intermittent Pemigatinib 1 mg QD | Part 1: Intermittent Pemigatinib 2 mg QD | Part 1: Intermittent Pemigatinib 4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Intermittent/Continuous Pemigatinib 20 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 18 | 57 | 13
ratio | 1.09 (NA) — A standard deviation was not calculated for a single participant. | 1.64 (NA) — A standard deviation was not calculated for a single participant. | 1.36 (NA) — A standard deviation was not calculated for a single participant. | 1.67 (0.264) | 1.71 (0.534) | 1.69 (0.538) | 1.76 (0.476)

21. Secondary Outcome: Parts 1 and 2: Cmax Steady State Following Administration of Pemigatinib in the Fasted (Cycle 1 Day 14) and Fed (Cycle 2 Day 14) States
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: Cycles 1 and 2: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Day 14
Population: PK/PD Population. Only participants who participated in the food-effect study in Part 2 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted: Participants self-administered intermittent or continuous pemigatinib 13.5 mg QD in the fasted state in Part 2. Intermittent dosing: participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. Continuous dosing: participants self-administered oral pemigatinib 13.5 mg QD on Days 1 through 21 of each 21-day cycle.
- Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed: Participants self-administered intermittent or continuous pemigatinib 13.5 mg QD in the fed state in Part 2. Intermittent dosing: participants self-administered oral pemigatinib 13.5 mg QD on a 2-weeks-on therapy and 1-week-off therapy schedule. The treatment cycle consisted of: Days 1 through 14: pemigatinib QD; Days 15 through 21: treatment break. Continuous dosing: participants self-administered oral pemigatinib 13.5 mg QD on Days 1 through 21 of each 21-day cycle.
Arm/Group | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed
Number analyzed (Participants) | 12 | 12
ng/mL | 215 (86.5) | 179 (82.8)
Statistical Analysis 1: Comparison: Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted vs Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed; Test type: Superiority; p = 0.143, ANOVA; crossover ANOVA of log-transformed data

22. Secondary Outcome: Parts 1 and 2: Tmax Steady State Following Administration of Pemigatinib in the Fasted (Cycle 1 Day 14) and Fed (Cycle 2 Day 14) States
Description: tmax was defined as the time to the maximum observed plasma concentration.
Time Frame: Cycles 1 and 2: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Day 14
Population: PK/PD Population. Only participants who participated in the food-effect study in Part 2 were analyzed.
Measure: Median (Full Range); unit: hr
Arm/Group | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed
Number analyzed (Participants) | 12 | 12
hr | 1.58 [0.500 to 5.78] | 4.02 [1.00 to 7.58]
Statistical Analysis 1: Comparison: Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted vs Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed; Test type: Superiority; p = 0.0013, ANOVA; crossover ANOVA of log-transformed data

23. Secondary Outcome: Parts 1 and 2: t1/2 Steady State Following Administration of Pemigatinib in the Fasted (Cycle 1 Day 14) and Fed (Cycle 2 Day 14) States
Description: t1/2 was defined as the apparent plasma terminal phase disposition half-life.
Time Frame: Cycles 1 and 2: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Day 14
Population: PK/PD Population. Only participants who participated in the food-effect study in Part 2 were analyzed.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed
Number analyzed (Participants) | 12 | 12
hr | 19.2 (10.5) | 23.8 (17.5)
Statistical Analysis 1: Comparison: Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted vs Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed; Test type: Superiority; p = 0.319, ANOVA; crossover ANOVA of log-transformed data

24. Secondary Outcome: Parts 1 and 2: Cmin Steady State Following Administration of Pemigatinib in the Fasted (Cycle 1 Day 14) and Fed (Cycle 2 Day 14) States
Description: Cmin was defined as the minimum observed plasma concentration over the dose interval.
Time Frame: Cycles 1 and 2: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Day 14
Population: PK/PD Population. Only participants who participated in the food-effect study in Part 2 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed
Number analyzed (Participants) | 12 | 12
ng/mL | 61.1 (33.5) | 65.7 (34.7)
Statistical Analysis 1: Comparison: Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted vs Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed; Test type: Superiority; p = 0.128, ANOVA; crossover ANOVA of log-transformed data

25. Secondary Outcome: Parts 1 and 2: AUC0-24 Steady State Following Administration of Pemigatinib in the Fasted (Cycle 1 Day 14) and Fed (Cycle 2 Day 14) States
Description: AUC0-24 was defined as the area under the plasma or serum concentration-time curve from time 0 to 24 hours post-dose.
Time Frame: Cycles 1 and 2: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Day 14
Population: PK/PD Population. Only participants who participated in the food-effect study in Part 2 were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 2580 (999) | 2910 (1310)
Statistical Analysis 1: Comparison: Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted vs Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed; Test type: Superiority; p = 0.305, ANOVA; crossover ANOVA of log-transformed data

26. Secondary Outcome: Parts 1 and 2: CL/F Steady State Following Administration of Pemigatinib in the Fasted (Cycle 1 Day 14) and Fed (Cycle 2 Day 14) States
Description: CL/F was defined as the apparent oral dose clearance.
Time Frame: Cycles 1 and 2: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Day 14
Population: PK/PD Population. Only participants who participated in the food-effect study in Part 2 were analyzed.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed
Number analyzed (Participants) | 12 | 12
L/hr | 12.4 (4.94) | 11.3 (4.87)
Statistical Analysis 1: Comparison: Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted vs Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed; Test type: Superiority; p = 0.305, ANOVA; crossover ANOVA of log-transformed data

27. Secondary Outcome: Parts 1 and 2: Vz/F Steady State Following Administration of Pemigatinib in the Fasted (Cycle 1 Day 14) and Fed (Cycle 2 Day 14) States
Description: Vz/F was defined as the apparent volume of distribution.
Time Frame: Cycles 1 and 2: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Day 14
Population: PK/PD Population. Only participants who participated in the food-effect study in Part 2 were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted | Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed
Number analyzed (Participants) | 12 | 12
Liters | 307 (139) | 364 (262)
Statistical Analysis 1: Comparison: Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fasted vs Part 2: Intermittent/Continuous Pemigatinib 13.5 mg QD, Fed; Test type: Superiority; p = 0.772, ANOVA; crossover ANOVA of log-transformed data

28. Secondary Outcome: Part 3: Cmax of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 1
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 1
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 19 | 7 | 7 | 6
ng/mL | 137 (65.7) | 199 (99.6) | 234 (84.1) | 214 (98.2) | 259 (55.4)

29. Secondary Outcome: Part 3: Tmax of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 1
Description: tmax was defined as the time to the maximum observed plasma concentration.
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 1
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: hr
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 19 | 7 | 7 | 6
hr | 1.98 [1.00 to 4.00] | 1.05 [0.500 to 23.4] | 2.00 [0.500 to 22.6] | 1.00 [0.500 to 3.98] | 0.783 [0.500 to 18.6]

30. Secondary Outcome: Part 3: AUClast of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 1
Description: as for outcome 11
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 1
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 19 | 7 | 7 | 6
hr*ng/mL | 1480 (587) | 1880 (821) | 2890 (1010) | 1890 (491) | 2040 (513)

31. Secondary Outcome: Part 3: AUC0-24 of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 1
Description: AUC0-24 was defined as the area under the plasma or serum concentration-time curve from time 0 to 24 hours post-dose.
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 1
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 19 | 7 | 7 | 6
hr*ng/mL | 1550 (552) | 1910 (838) | 2920 (1070) | 1890 (471) | 1890 (269)

32. Secondary Outcome: Part 3: Cmax of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 14 (Steady State)
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 14
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 14 | 4 | 5 | 5
ng/mL | 166 (52.1) | 255 (119) | 214 (203) | 231 (99.4) | 404 (41.7)

33. Secondary Outcome: Part 3: Tmax of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 14 (Steady State)
Description: tmax was defined as the time to the maximum observed plasma concentration.
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 14
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: hr
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 14 | 4 | 5 | 5
hr | 5.78 [1.25 to 6.08] | 1.08 [0.500 to 7.98] | 1.50 [0.950 to 4.00] | 1.90 [0.500 to 2.08] | 0.583 [0.500 to 1.07]

34. Secondary Outcome: Part 3: t1/2 of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 14 (Steady State)
Description: t1/2 was defined as the apparent plasma terminal phase disposition half-life.
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 14
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 14 | 4 | 5 | 5
hr | 15.3 (0.207) | 17.0 (6.90) | 10.6 (3.29) | 14.7 (6.43) | 15.3 (2.64)

35. Secondary Outcome: Part 3: Cmin of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 14 (Steady State)
Description: Cmin was defined as the minimum observed plasma concentration over the dose interval.
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 14
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 14 | 4 | 5 | 5
ng/mL | 58.0 (31.6) | 56.6 (31.3) | 48.5 (57.8) | 63.1 (32.4) | 64.2 (25.8)

36. Secondary Outcome: Part 3: AUC0-24 of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 14 (Steady State)
Description: AUC0-24 was defined as the area under the plasma or serum concentration-time curve from time 0 to 24 hours post-dose.
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 14
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 14 | 4 | 5 | 5
hr*ng/mL | 2400 (628) | 2400 (967) | 1650 (1060) | 2910 (1390) | 3440 (672)

37. Secondary Outcome: Part 3: CL/F of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 14 (Steady State)
Description: CL/F was defined as the apparent oral dose clearance.
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 14
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 14 | 4 | 5 | 5
L/hr | 8.03 (1.89) | 13.4 (5.46) | 24.5 (17.7) | 12.7 (9.03) | 8.26 (1.39)

38. Secondary Outcome: Part 3: Vz/F of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 14 (Steady State)
Description: Vz/F was defined as the apparent volume of distribution.
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 14
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 14 | 4 | 5 | 5
Liters | 177 (39.8) | 303 (136) | 376 (261) | 227 (82.2) | 182 (43.2)

39. Secondary Outcome: Part 3: Accumulation Ratio of Pemigatinib as Part of Combination Therapy on Cycle 1 Day 14 (Steady State)
Description: as for outcome 20
Time Frame: predose and 0.5, 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 14
Population: PK/PD Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg
Number analyzed (Participants) | 3 | 14 | 4 | 5 | 5
ratio | 1.65 (0.501) | 1.53 (0.381) | 0.604 (0.265) | 1.52 (0.772) | 1.90 (0.432)

ADVERSE EVENTS:
Time Frame: up to 869 days
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug and within 30 days of the last dose of study drug, are reported for all enrolled participants who received at least 1 dose of study drug (Safety Population).
Arm/Group | Part 1: Intermittent Pemigatinib 1/2/4 mg QD | Part 1: Intermittent Pemigatinib 6 mg QD | Parts 1 and 2: Intermittent Pemigatinib 9 mg QD | Parts 1 and 2: Intermittent Pemigatinib 13.5 mg QD | Part 1: Intermittent Pemigatinib 20 mg QD | Parts 1 and 2: Continuous Pemigatinib 9 mg QD | Parts 1 and 2: Continuous Pemigatinib 13.5 mg QD | Parts 1 and 2: Continuous Pemigatinib 20 mg QD | Part 1: Continuous Pemigatinib 7.5 mg BID | Part 1: Continuous Pemigatinib 10 mg BID | Part 3: Gem/Cis/Intermittent Pemigatinib 9 mg | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg | Part 3: Tras/Intermittent Pemigatinib 13.5 mg | Part 3: Doc/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Intermittent Pemigatinib 9 mg | Part 3: Pem/Intermittent Pemigatinib 13.5 mg | Part 3: Pem/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 9 mg | Part 3: Ref/Continuous Pemigatinib 13.5 mg | Part 3: Ref/Continuous Pemigatinib 20 mg
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/4 | 6/7 | 37/50 | 6/6 | 10/14 | 21/30 | 10/15 | 4/4 | 2/3 | 1/1 | 7/7 | 5/6 | 5/7 | 3/3 | 9/14 | 6/9 | 6/7 | 3/9 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4 | 3/7 | 21/50 | 3/6 | 6/14 | 14/30 | 7/15 | 2/4 | 2/3 | 1/1 | 3/7 | 0/6 | 6/7 | 1/3 | 7/14 | 3/9 | 4/7 | 5/9 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 7/7 | 50/50 | 6/6 | 14/14 | 30/30 | 15/15 | 4/4 | 3/3 | 1/1 | 7/7 | 6/6 | 7/7 | 3/3 | 14/14 | 9/9 | 7/7 | 9/9 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Intermittent Pemigatinib 1/2/4 mg QD (N=3) | Part 1: Intermittent Pemigatinib 6 mg QD (N=4) | Parts 1 and 2: Intermittent Pemigatinib 9 mg QD (N=7) | Parts 1 and 2: Intermittent Pemigatinib 13.5 mg QD (N=50) | Part 1: Intermittent Pemigatinib 20 mg QD (N=6) | Parts 1 and 2: Continuous Pemigatinib 9 mg QD (N=14) | Parts 1 and 2: Continuous Pemigatinib 13.5 mg QD (N=30) | Parts 1 and 2: Continuous Pemigatinib 20 mg QD (N=15) | Part 1: Continuous Pemigatinib 7.5 mg BID (N=4) | Part 1: Continuous Pemigatinib 10 mg BID (N=3) | Part 3: Gem/Cis/Intermittent Pemigatinib 9 mg (N=1) | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg (N=7) | Part 3: Tras/Intermittent Pemigatinib 13.5 mg (N=6) | Part 3: Doc/Intermittent Pemigatinib 13.5 mg (N=7) | Part 3: Pem/Intermittent Pemigatinib 9 mg (N=3) | Part 3: Pem/Intermittent Pemigatinib 13.5 mg (N=14) | Part 3: Pem/Continuous Pemigatinib 13.5 mg (N=9) | Part 3: Ref/Continuous Pemigatinib 9 mg (N=7) | Part 3: Ref/Continuous Pemigatinib 13.5 mg (N=9) | Part 3: Ref/Continuous Pemigatinib 20 mg (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood osmolarity decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin I (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Intermittent Pemigatinib 1/2/4 mg QD (N=3) | Part 1: Intermittent Pemigatinib 6 mg QD (N=4) | Parts 1 and 2: Intermittent Pemigatinib 9 mg QD (N=7) | Parts 1 and 2: Intermittent Pemigatinib 13.5 mg QD (N=50) | Part 1: Intermittent Pemigatinib 20 mg QD (N=6) | Parts 1 and 2: Continuous Pemigatinib 9 mg QD (N=14) | Parts 1 and 2: Continuous Pemigatinib 13.5 mg QD (N=30) | Parts 1 and 2: Continuous Pemigatinib 20 mg QD (N=15) | Part 1: Continuous Pemigatinib 7.5 mg BID (N=4) | Part 1: Continuous Pemigatinib 10 mg BID (N=3) | Part 3: Gem/Cis/Intermittent Pemigatinib 9 mg (N=1) | Part 3: Gem/Cis/Intermittent Pemigatinib 13.5 mg (N=7) | Part 3: Tras/Intermittent Pemigatinib 13.5 mg (N=6) | Part 3: Doc/Intermittent Pemigatinib 13.5 mg (N=7) | Part 3: Pem/Intermittent Pemigatinib 9 mg (N=3) | Part 3: Pem/Intermittent Pemigatinib 13.5 mg (N=14) | Part 3: Pem/Continuous Pemigatinib 13.5 mg (N=9) | Part 3: Ref/Continuous Pemigatinib 9 mg (N=7) | Part 3: Ref/Continuous Pemigatinib 13.5 mg (N=9) | Part 3: Ref/Continuous Pemigatinib 20 mg (N=2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 10 (10) | 1 (1) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (7) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 4 (6) | 0 (0) | 5 (5) | 7 (11) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (10) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 15 (15) | 1 (1) | 6 (7) | 11 (12) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 3 (4) | 0 (0) | 6 (6) | 5 (5) | 1 (1) | 3 (3) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 10 (14) | 2 (2) | 6 (8) | 6 (9) | 4 (5) | 2 (3) | 1 (1) | 1 (1) | 7 (8) | 2 (2) | 3 (3) | 1 (1) | 7 (10) | 3 (4) | 2 (2) | 0 (0) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 4 (5) | 4 (6) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (7) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 7 (8) | 0 (0) | 5 (5) | 7 (10) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (9) | 1 (1) | 0 (0) | 0 (0) | 5 (10) | 3 (4) | 0 (0) | 2 (4) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood 1,25-dihydroxycholecalciferol decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood 1,25-dihydroxycholecalciferol increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood 25-hydroxycholecalciferol decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 5 (7) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (5) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 11 (18) | 4 (4) | 1 (4) | 0 (0) | 1 (1) | 4 (6) | 1 (1) | 1 (1) | 1 (1) | 4 (7) | 1 (1) | 1 (2) | 2 (5) | 2 (4)
Blood folate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast fibrosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract cortical (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Computerised tomogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 14 (14) | 2 (2) | 4 (4) | 12 (13) | 4 (6) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 3 (4) | 0 (0) | 5 (7) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal epithelium defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 12 (12) | 1 (1) | 1 (1) | 11 (11) | 5 (5) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (2) | 0 (0) | 9 (11) | 2 (2) | 1 (1) | 3 (6) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (7) | 1 (2) | 1 (1) | 4 (4) | 4 (4) | 4 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (7) | 1 (1) | 2 (3) | 1 (1) | 3 (3) | 3 (6) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3) | 12 (12) | 2 (2) | 3 (3) | 15 (18) | 9 (12) | 1 (2) | 1 (2) | 0 (0) | 4 (7) | 3 (3) | 6 (13) | 1 (1) | 7 (17) | 3 (7) | 3 (6) | 3 (6) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 1 (1) | 1 (2) | 10 (11) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (5) | 17 (19) | 2 (2) | 5 (5) | 13 (13) | 8 (8) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 4 (5) | 5 (5) | 4 (4) | 3 (3) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 9 (9) | 4 (5) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Entropion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 1 (1) | 1 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (3) | 5 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 4 (4) | 18 (21) | 2 (2) | 8 (8) | 8 (8) | 4 (5) | 2 (3) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 5 (6) | 1 (1) | 5 (5) | 1 (1) | 3 (3) | 6 (10) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Growth of eyelashes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (8) | 0 (0) | 2 (2) | 8 (9) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism secondary (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 4 (13) | 39 (78) | 4 (6) | 8 (12) | 28 (49) | 13 (19) | 4 (5) | 3 (5) | 1 (1) | 3 (6) | 5 (9) | 6 (7) | 3 (4) | 11 (41) | 5 (7) | 4 (4) | 5 (9) | 2 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 1 (2) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 0 (0) | 8 (14) | 4 (5) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4) | 10 (17) | 1 (1) | 0 (0) | 5 (7) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation decreased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 7 (7) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 8 (8) | 2 (2) | 6 (6) | 13 (15) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 4 (6) | 0 (0) | 3 (8) | 3 (3) | 2 (4) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (9) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular surface disease (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oesophageal hypomotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 9 (11) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 6 (7) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 7 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 0 (0) | 4 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 5 (6) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (1) | 8 (9) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 2 (3) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic pemphigus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (4) | 4 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal fovea disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral discolouration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Steroid withdrawal syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 11 (13) | 3 (3) | 6 (8) | 15 (18) | 7 (11) | 2 (2) | 3 (5) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 5 (7) | 3 (4) | 4 (5) | 7 (10) | 1 (1)
Subretinal fluid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichiasis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 3 (5) | 2 (4) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 5 (5) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 7 (7) | 1 (1) | 4 (4) | 9 (12) | 3 (6) | 2 (4) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 3 (5) | 1 (1) | 3 (5) | 3 (3) | 2 (4) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 3 (3) | 3 (3) | 5 (7) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT02393248/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT02393248/SAP_001.pdf